CLINICAL TRIAL: NCT01136577
Title: Comparison of Light-emitting Diodes (LED) Phototherapy Versus Fluorescent Lamps Phototherapy for Treatment of Hyperbilirubinemia in Term Newborn
Brief Title: Light-emitting Diodes (LED) Phototherapy for Hyperbilirubinemia of Term Newborn
Acronym: DELF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070604
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Hyperbilirubinemia
Keywords: Jaundice; Hyperbilirubinemia; Phototherapy; term newborn; LED; Fluorescent lamps
MeSH Terms: conditions — Hyperbilirubinemia; Jaundice | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LEDDYBLOO® (Experimental): LEDDYBLOO® phototherapy device equipped with 20 at 30 blue and white LEDs
  Interventions: Device: Phototherapy
- Double BILITRON® (Experimental): Double BILITRON® phototherapy corresponding to two small ramps associated together each one equipped of 5 blue LEDS
  Interventions: Device: Phototherapy
- Futura® (Experimental): Future phototherapy device equipped with 8 fluorescent tubes
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy — Phototherapy devices of ramp type placed over the incubator to treat with light in the 420-490nm range one face of the naked baby suffering jaundice.

SUMMARY:
Phototherapy is almost (beside exchange transfusion) the unique treatment for hyperbilirubinemia of the newborn. Its efficacy to decrease bilirubin level (because the light interacts with bilirubin at the skin level to transform it in water soluble products eliminated in urine and stools without liver metabolism) relies on the irradiance dispensed at the skin level by the device (in the 430-490nm range) and on the exposed surface of the baby. In the past years, technology of phototherapy devices moved from fluorescent lamps to LED, improving the amount of light energy emitted but on a smaller surface. The purpose of the study is to compare the efficacy of three ramps of phototherapy, one equipped with fluorescent tubes and two with LED (in a different technological settings) in the treatment of term (35 GW or more) healthy newborn suffering hyperbilirubinemia after 2days of life.

DETAILED DESCRIPTION:
Term and healthy newborns on maternity wards in SAINT-ANTOINE hospital are checked everyday for jaundice with bilirubinometer JM-103®. If indicated (nomogram included in patient charts), a plasmatic bilirubin level is performed. If the baby is two days old or more with a bilirubin level indicating standard phototherapy (by opposition to intensive phototherapy), the parents are informed of the research protocol and after obtention of parental consent, the baby is included. The newborn is admitted in the neonatology unit and randomised in one of the three phototherapy devices group. Plasmatic bilirubin levels are checked at 6,12 and 24 and 48 hours of phototherapy. At 12 hours of phototherapy, a biological checking is performed to address the etiology of the jaundice. The next plasmatic bilirubin level is performed at 72h after inclusion. During phototherapy treatment the baby is continuously monitored. Phototherapy is stopped when bilirubin level is below 200µmol/l. If the bilirubin level is increasing under one of this ramps or does not decrease at H24, the baby will be immediately move on intensive phototherapy and participation at the research protocol interrupted. Twenty four hours after the end of phototherapy treatment, plasmatic bilirubin level is checked to confirm the end of jaundice and statement is made for jaundice origin. The total duration of participation of a baby at this study is 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Newborns in the hospital SAINT ANTOINE maternity wards
* Gestational age of 35w or more
* Healthy (no hypoxemia, no hypotonia, no abnormalities of thermic regulation, no infection or dehydration)
* No foeto-maternal incompatibility in rhesus or kell group
* With bilirubin level at 48h of 220µmoles/l or more if born at 38W or more or of 200µmoles/l or more if born between 35 and 38 W
* Parental information done and signed consent obtained
* Parents affiliated to social security

Exclusion Criteria:

* Conjugated bilirubin level at 25µmol/l or more
* Total bilirubin level over 300µmol/l indicating "intensive phototherapy"
* Baby treated by phototherapy in the days before inclusion
* Severe haemolytic disease with anemia below 14g/land or hyperbilirubinemia before 48h of life), rhesus or kell incompatibility
* Parents who could not understand the information or sign the consent.

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Bilirubinemia | 24 hours

SECONDARY OUTCOMES:
Evolution of bilirubinemia according to the device used | 6, 12,24, 48, 72 hours
Hyperbilirubinemia rebound according to the device used | 24 and 48 hours after discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Anne Cortey, Doctor, Principal Investigator — APHP
Locations (1):
- CNRHP, Saint Antoine Hospital, Paris, France, France

REFERENCES:
- [Background] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951
- [Background] Bertini G, Dani C, Pezzati M, Rubaltelli FF. Prevention of bilirubin encephalopathy. Biol Neonate. 2001;79(3-4):219-23. doi: 10.1159/000047095. PMID 11275655
- [Background] Bertini G, Perugi S, Elia S, Pratesi S, Dani C, Rubaltelli FF. Transepidermal water loss and cerebral hemodynamics in preterm infants: conventional versus LED phototherapy. Eur J Pediatr. 2008 Jan;167(1):37-42. doi: 10.1007/s00431-007-0421-3. Epub 2007 Feb 13. PMID 17297614
- [Background] Bertini G, Dani C, Tronchin M, Rubaltelli FF. Is breastfeeding really favoring early neonatal jaundice? Pediatrics. 2001 Mar;107(3):E41. doi: 10.1542/peds.107.3.e41. PMID 11230622
- [Background] Bhutani VK, Johnson L, Sivieri EM. Predictive ability of a predischarge hour-specific serum bilirubin for subsequent significant hyperbilirubinemia in healthy term and near-term newborns. Pediatrics. 1999 Jan;103(1):6-14. doi: 10.1542/peds.103.1.6. PMID 9917432
- [Background] Bhutani VK, Johnson L. Prevention of severe neonatal hyperbilirubinemia in healthy infants of 35 or more weeks of gestation: implementation of a systems-based approach. J Pediatr (Rio J). 2007 Jul-Aug;83(4):289-93. doi: 10.2223/JPED.1673. No abstract available. PMID 17676232
- [Background] Bhutani VK, Maisels MJ, Stark AR, Buonocore G; Expert Committee for Severe Neonatal Hyperbilirubinemia; European Society for Pediatric Research; American Academy of Pediatrics. Management of jaundice and prevention of severe neonatal hyperbilirubinemia in infants >or=35 weeks gestation. Neonatology. 2008;94(1):63-7. doi: 10.1159/000113463. Epub 2008 Jan 17. PMID 18204221
- [Background] Bhutani VK, Johnson LH, Keren R. Diagnosis and management of hyperbilirubinemia in the term neonate: for a safer first week. Pediatr Clin North Am. 2004 Aug;51(4):843-61, vii. doi: 10.1016/j.pcl.2004.03.011. PMID 15275978
- [Background] Chang YS, Hwang JH, Kwon HN, Choi CW, Ko SY, Park WS, Shin SM, Lee M. In vitro and in vivo efficacy of new blue light emitting diode phototherapy compared to conventional halogen quartz phototherapy for neonatal jaundice. J Korean Med Sci. 2005 Feb;20(1):61-4. doi: 10.3346/jkms.2005.20.1.61. PMID 15716604
- [Background] Cohen SM. Jaundice in the full-term newborn. Pediatr Nurs. 2006 May-Jun;32(3):202-8. PMID 16802676
- [Background] Grohmann K, Roser M, Rolinski B, Kadow I, Muller C, Goerlach-Graw A, Nauck M, Kuster H. Bilirubin measurement for neonates: comparison of 9 frequently used methods. Pediatrics. 2006 Apr;117(4):1174-83. doi: 10.1542/peds.2005-0590. PMID 16585313
- [Background] Hansen TW. Acute management of extreme neonatal jaundice--the potential benefits of intensified phototherapy and interruption of enterohepatic bilirubin circulation. Acta Paediatr. 1997 Aug;86(8):843-6. doi: 10.1111/j.1651-2227.1997.tb08608.x. PMID 9307164
- [Background] Lindgren C, Nilsson T. [Treatment of neonatal hyperbilirubinemia with BiliBed]. Tidsskr Nor Laegeforen. 1999 Nov 10;119(27):4027-9. Norwegian. PMID 10613092
- [Background] Maisels MJ, Kring E. Transcutaneous bilirubin levels in the first 96 hours in a normal newborn population of > or = 35 weeks' gestation. Pediatrics. 2006 Apr;117(4):1169-73. doi: 10.1542/peds.2005-0744. PMID 16585312
- [Background] Maisels MJ. What's in a name? Physiologic and pathologic jaundice: the conundrum of defining normal bilirubin levels in the newborn. Pediatrics. 2006 Aug;118(2):805-7. doi: 10.1542/peds.2006-0675. No abstract available. PMID 16882840
- [Background] Maisels MJ, McDonagh AF. Phototherapy for neonatal jaundice. N Engl J Med. 2008 Feb 28;358(9):920-8. doi: 10.1056/NEJMct0708376. No abstract available. PMID 18305267
- [Background] Maisels MJ, Newman TB. Surveillance of severe neonatal hyperbilirubinemia: a view from south of the border. CMAJ. 2006 Sep 12;175(6):599. doi: 10.1503/cmaj.060960. No abstract available. PMID 16966662
- [Background] Newman TB, Liljestrand P, Jeremy RJ, Ferriero DM, Wu YW, Hudes ES, Escobar GJ; Jaundice and Infant Feeding Study Team. Outcomes among newborns with total serum bilirubin levels of 25 mg per deciliter or more. N Engl J Med. 2006 May 4;354(18):1889-900. doi: 10.1056/NEJMoa054244. PMID 16672700
- [Background] Newman TB, Liljestrand P, Escobar GJ. Combining clinical risk factors with serum bilirubin levels to predict hyperbilirubinemia in newborns. Arch Pediatr Adolesc Med. 2005 Feb;159(2):113-9. doi: 10.1001/archpedi.159.2.113. PMID 15699303
- [Background] Rubaltelli FF, Gourley GR, Loskamp N, Modi N, Roth-Kleiner M, Sender A, Vert P. Transcutaneous bilirubin measurement: a multicenter evaluation of a new device. Pediatrics. 2001 Jun;107(6):1264-71. doi: 10.1542/peds.107.6.1264. PMID 11389241
- [Background] Seidman DS, Moise J, Ergaz Z, Laor A, Vreman HJ, Stevenson DK, Gale R. A new blue light-emitting phototherapy device: a prospective randomized controlled study. J Pediatr. 2000 Jun;136(6):771-4. PMID 10839875
- [Background] Seidman DS, Moise J, Ergaz Z, Laor A, Vreman HJ, Stevenson DK, Gale R. A prospective randomized controlled study of phototherapy using blue and blue-green light-emitting devices, and conventional halogen-quartz phototherapy. J Perinatol. 2003 Mar;23(2):123-7. doi: 10.1038/sj.jp.7210862. PMID 12673261
- [Background] Shapiro SM. Bilirubin toxicity in the developing nervous system. Pediatr Neurol. 2003 Nov;29(5):410-21. doi: 10.1016/j.pediatrneurol.2003.09.011. PMID 14684236
- [Background] Smitherman H, Stark AR, Bhutani VK. Early recognition of neonatal hyperbilirubinemia and its emergent management. Semin Fetal Neonatal Med. 2006 Jun;11(3):214-24. doi: 10.1016/j.siny.2006.02.002. PMID 16603425
- [Background] Stokowski LA. Fundamentals of phototherapy for neonatal jaundice. Adv Neonatal Care. 2006 Dec;6(6):303-12. doi: 10.1016/j.adnc.2006.08.004. PMID 17208161